CLINICAL TRIAL: NCT00002156
Title: A Randomized Comparison of Intravitreal ISIS 2922 Plus Ganciclovir Versus Ganciclovir as Treatment for Patients With Cytomegalovirus Retinitis ( CMVR )
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 251B; ISIS 2922-CS3
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiviral Agents; Cytomegalovirus Retinitis; Injections
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — fomivirsen; Ganciclovir

INTERVENTIONS:
Drug: Fomivirsen sodium
Drug: Ganciclovir

SUMMARY:
To determine the clinically safe and effective dose of intravitreal ISIS 2922 alone and as an additive antiviral therapy to ganciclovir in AIDS patients with cytomegalovirus (CMV) retinitis.

DETAILED DESCRIPTION:
In Stage 1 of the study, 20 patients receive one of two doses of ISIS 2922 on days 1, 8, and 15 (Induction) then every 14 days (maintenance), with ganciclovir given daily during both Induction and Maintenance. Escalation to the second dose does not occur until all patients at the first dose level have reached their first maintenance dose (day 29). In Stage 2 of the study, 174 patients are randomized to receive either a) ISIS 2922 at the dose established in Stage 1 on days 1, 8, and 15 and then every 14 days, with ganciclovir given daily during both Induction and Maintenance, or b) ganciclovir daily for 14 consecutive days and then a lower dose as maintenance. Patients may continue to receive ISIS 2922 biweekly if the dose is safe and their CMV retinitis is clinically controlled. Per 2/8/96 amendment, patients are now in Stage 2 at 150 mcg.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS.
* CMV retinitis that is not adequately controlled (previously diagnosed patients with smoldering CMV retinitis or those with active CMV retinitis borders on indirect ophthalmoscopy).
* No more than one previous progression of CMV retinitis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions in the eye to be treated are excluded:

* External ocular infection.
* Other herpetic infections of the retina, toxoplasma retinochoroiditis, or other disease of the fundus.
* Ocular condition that will obstruct visualization of the posterior ocular structures.
* Retinal detachment.
* Silicone oil in eye.

Patients with the following other symptoms or conditions are excluded:

* Known or suspected allergy to phosphorothioate oligonucleotides.
* Syphilis.
* Retinal pigment epithelial stippling not associated with CMV retinitis.
* Pseudoretinitis pigmentosa.
* Chronic diarrhea that would impair absorption of oral ganciclovir.
* Intolerance to ganciclovir.

Concurrent Medication:

Excluded:

* Foscarnet or other anti-CMV agents other than ganciclovir.
* Mellaril.
* Stelazine.
* Thorazine.
* Clofazimine.
* Ethambutol/fluconazole combination.
* Investigational medications for CMV retinitis.

Concurrent Treatment:

Excluded:

* Investigational procedures for CMV retinitis.

Patients with the following prior conditions are excluded:

* History of surgery to correct retinal detachment in eye to be treated.
* History of intolerance to ISIS 2922.

Prior Medication:

Excluded:

* Prior ganciclovir implant for CMV retinitis.
* More than 4 months of prior ganciclovir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Retina - Vitreous Associates Med Group, Los Angeles, California
  - Community Eye Med Group, Pasadena, California
  - San Diego Naval Hosp, San Diego, California
  - Univ of California San Francisco / SF Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Dr Julio Perez, Fort Lauderdale, Florida
  - Georgia Retina, Atlanta, Georgia
  - Univ of Illinois, Chicago, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - Vitreo - Retinal Consultants, New York, New York
  - Charlotte Eye Ear Nose and Throat Association, Charlotte, North Carolina
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Novum Inc, Seattle, Washington